CLINICAL TRIAL: NCT06374953
Title: A Novel Viscoelastic Test Based on Ultrasonic Guided Wave for Identifying Hyperfibrinolysis Rapidly
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0182
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-03

CONDITIONS: Hyperfibrinolysis
Keywords: fibrinolysis; blood coagulation tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound-based viscoelastic hemostasis analysis — Adding recombinant tissue plasminogen activator (rtPA) and/or Tranexamic acid （TXA）to blood in vitro, and fibrinolysis capacity is assessed using ultrasound-guided viscoelastic coagulation testing.

SUMMARY:
This study compares the results of the existing fibrinolysis monitoring technology to the Ultrasound-based viscoelastic hemostasis analysis, a new method, using small amount of extra blood obtained during routine blood draws in surgery patients.

DETAILED DESCRIPTION:
Ultrasound-based viscoelastic hemostasis analysis is a novel POC diagnostic method, which is suitable for operating theatres and emergency rooms.

The novel viscoelastic hemostasis analysis uses ultrasound guided waves to characterize the dynamic changes in viscoelastic properties of a blood sample during coagulation and clot lysis, which will be an assay of hyperfibrinolysis for critically ill patients.

This single-center, prospective, observational pilot study will evaluate the analytical performance as well as compared to conventional viscoelastic testing methods.

ELIGIBILITY:
PART 1

Inclusion Criteria:

Subject is scheduled for surgery with general surgery Subject is 18 years or order Subject requires routine TEG measurement

Exclusion Criteria:

Subject with coagulation and fibrinolysis exceeding normal values based on laboratory tests (including prothrombin time, international normalized ratio, activated partial thromboplastin time, plasma fibrinogen concentration, D-dimer, platelet count, hemoglobin concentration, and hematocrit) Subject with any abnormal parameters detected by TEG Subject with a history of bleeding and thrombosis Subject who has taken any medications that may affect coagulation, platelet aggregation, or fibrinolysis within the past 10 days (including non-steroidal anti-inflammatory drugs and aspirin) Residual blood volume <1ml

PART 2

Inclusion Criteria:

Subject is scheduled for surgery with general surgery Subject is 18 years or order Subject Subjects with detected hyperfibrinolysis (LY30>8%) or non-hyperfibrinolysis(LY30≤8%) based on TEG.

Exclusion Criteria:

Residual blood volume <1ml

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants for this study will be recruited at the Second Affiliated Hospital Zhejiang University School of Medicine. The study participants will be adult general anesthesia patients with viscoelastic testing performed to assess fibrinolysis.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of the novel viscoelastic hemostasis analysis results to TEG-LY30 | 1 day
  Fibrinolysis capacity assessed by the novel viscoelastic hemostasis analysis and TEG-LY30

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University anesthesiology department, Hangzhou, Zhejiang, China